CLINICAL TRIAL: NCT05431946
Title: Palliative Care for Patients With Liver Cirrhosis - a Multicentre Intervention Study
Brief Title: Palliative Care for Patients With Liver Cirrhosis
Acronym: LiverCare
Status: Enrolling by invitation | Type: Observational
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Collaborators: Herlev Hospital (Other); Aarhus University Hospital (Other); Hvidovre University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LiverCare Denmark
Record Dates: First submitted 2022-05-11; First posted 2022-06-24 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: End of Life Care; Liver Cirrhosis; Nurse-Patient Relations; Quality of Life
MeSH Terms: conditions — Liver Cirrhosis | interventions — Advance Care Planning; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Palliative Care arm: Intervention by Advance care planning (ACP) conversation:The goal is the identification, assessment, and treatment of physical, psychosocial, or spiritual symptoms and problems.
  Advance care actions:These are the actions taken to fulfill the advance care plan and can include, but are not limited to:treatments: pharmacological, psychosocial (priest, psychologist, etc.) referrals: rehabilitation, specialized palliative care team, hospice, etc.
  communication initiatives with relatives, primary care, public authorities
  Interventions: Behavioral: Advance Care Planning and the consequent actions
- Non-participating arm: Will continue standard of care

INTERVENTIONS:
Behavioral: Advance Care Planning and the consequent actions — The palliative care intervention is based on the advance care planning process and the actions taken as a consequence of these conversations. The goal is the identification, assessment, and treatment of physical, psychosocial, or spiritual symptoms and problems.
  Advance care actions
  These are the actions taken to fulfill the advance care plan and can include, but are not limited to:
  treatments: pharmacological, psychosocial (priest, psychologist, etc.) referrals: rehabilitation, specialized palliative care team, hospice, etc. communication initiatives with relatives, primary care, public authorities
  Other Names: Questionnaires
  Groups: Palliative Care arm

SUMMARY:
Background: Patients with liver cirrhosis rarely receive palliative care although the Danish Health Authorities and WHO recommend it. The lacking palliative intervention is probably owed to a physician culture focused on life-prolonging active treatment at any cost and unclarities, and misperceptions about palliative care, which is perceived by many as exclusively for cancer patients and something that marks the end of active treatment.

Study aim: Measure the effect of palliative care on the patient burden, caregiver burden, and the utilization of healthcare services.

Study design: Prospective multi-center intervention study with end of study at the patients' death. We will use a 3-faceted endpoint 1) Patient burden measured by change in Hospital Anxiety and Depression Scale, 2) caregiver burden by a change in Zarit Caregiver Burden Questionnaire, and 1) health care system burden as the difference in number, length, and indication for hospital admissions and need for outpatient services.

Patients: We will prospectively include 200 patients with liver cirrhosis (approx. 50 from each of 4-5 sites: Esbjerg, Herlev, Hvidovre, Århus) who have 2 or more items checked on the Supportive and Palliative Care Indicators Tool. Control groups will be identified from two non-participating hospitals and matched regarding age, gender, number of comorbidities, and alcohol and caregiver status.

Methods: The intervention will be advanced care planning with conversations and actions built around a standardized symptom identification tool (EORTC QLQ-C15-PAL). Advance care planning is the collaborative process between patients and health care professionals of planning future health care. The assignment of a contact nurse to each participant is a key part of the intervention.

Results: We will measure patient and caregiver burden at inclusion, after 4-6 weeks, 4-6 months, and every 6 months until the patient dies. All use of health care services will be registered. The use of health care services during the terminal 2 years will be compared that of control patients.

ELIGIBILITY:
Inclusion Criteria:

1. Liver cirrhosis of any etiology (diagnosed clinically, by imaging or histological features) as predominant chronic illness
2. 2 or more items checked on the Supportive and Palliative Care Indicators Tool (SPICT™, appendix)
3. Expressed desire for palliative support from the patient and relatives
4. Ability to give informed consent

Exclusion Criteria:

1. Inability to give informed consent
2. Age < 18 years
3. Ongoing contact with specialized palliative care teams or hospice
4. Other chronic life-threatening illness than liver cirrhosis is more likely to become the cause of death within 1-2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver cirrhosis
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Intra-subject change in patient burden | From date of inclusion until the date of death from any cause, assessed up to 100 months
  Change in Hospital Anxiety and Depression Scale

SECONDARY OUTCOMES:
Intra-subject change in caregiver burden | From date of inclusion until the date of death from any cause, assessed up to 100 months
  Change in Zarit Caregiver Burden Questionnaire
Inter-group difference in health care system burden | From date of inclusion until the date of death from any cause, assessed up to 100 months
  The difference in the use of health care services between intervention and control groups from 2 non-participating hospitals. The difference will be assessed by a review of electronic patient files and sundhed.dk.

CONTACTS AND LOCATIONS:
Overall Officials: Mette M Lauridsen, Principal Investigator — Head of Liver Research
Locations (1):
- Hospital of South West Jutland, Esbjerg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided